CLINICAL TRIAL: NCT03654729
Title: A Phase 3, Double-blind, Multicenter, Placebo-controlled Study of PledOx Used on Top of Modified FOLFOX6 (5-FU/FA and Oxaliplatin) to Prevent Chemotherapy Induced Peripheral Neuropathy (CIPN) in Patients With First-line mCRC
Brief Title: Preventive Treatment of Oxaliplatin Induced Peripheral Neuropathy in Metastatic Colorectal Cancer (POLAR-M)
Acronym: POLAR-M
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: On 23 January 2020, the Sponsor announced that the United States (US) Food and Drug Administration (FDA) had issued a clinical hold in the US of the POLAR program.
Sponsor: Egetis Therapeutics (Industry)
Collaborators: Solasia Pharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PP06490
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer; Chemotherapy-induced Peripheral Neuropathy
Keywords: Metastatic; Colorectal; Cancer; Metastatic Colorectal Cancer; Oxaliplatin induced CIPN; CIPN; Oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, multicenter, double-blind, placebo-controlled study to establish the efficacious dose of PledOx in prevention of chronic chemotherapy induced peripheral neuropathy (CIPN) induced by oxaliplatin.
  Patients with metastatic colorectal cancer (mCRC), who are indicated for first-line modified FOLFOX6 (mFOLFOX6) chemotherapy for at least 3 months, without any pre-planned treatment breaks, will be randomized in a 1:1:1 ratio, stratified by region (Asia, non-Asia) and PK sub-study (yes, no) to one of three treatment arms:
  * Arm A: PledOx (2 µmol/kg) + mFOLFOX6 chemotherapy
  * Arm B: PledOx (5 µmol/kg) + m
  * Arm C: Placebo + mFOLFOX6 chemotherapy
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PledOx (2 µmol/kg) (Experimental): Calmangafodipir (2 µmol/kg) on day 1 every two weeks to patients as an intravenous infusion, combined with mFOLFOX6 chemotherapy.
  Interventions: Drug: Calmangafodipir (2 µmol/kg)
- PledOx (5 µmol/kg) (Experimental): Calmangafodipir (5 µmol/kg) on day 1 every two weeks to patients as an intravenous infusion, combined with mFOLFOX6 chemotherapy.
  Interventions: Drug: Calmangafodipir (5 µmol/kg)
- Placebo (Placebo Comparator): Placebo will be given to patients as an intravenous infusion, on top of mFOLFOX6 chemotherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calmangafodipir (2 µmol/kg) — Solution in 20 mL single dose glass vials
  Other Names: PledOx
  Arms: PledOx (2 µmol/kg)
Drug: Calmangafodipir (5 µmol/kg) — Solution in 20 mL single dose glass vials
  Other Names: PledOx
  Arms: PledOx (5 µmol/kg)
Drug: Placebo — Solution in 20 mL single dose glass vials
  Arms: Placebo

SUMMARY:
This study evaluates the investigational drug PledOx in the prevention of chronic chemotherapy induced peripheral neuropathy (CIPN) induced by the drug oxaliplatin.

DETAILED DESCRIPTION:
Oxaliplatin, in combination with 5-fluorouracil plus folinate (or capecitabine), has increased survival in stage III colorectal cancer and prolonged life in stage IV patients, but its use is compromised because of severe toxicity. Chemotherapy-induced peripheral neuropathy (CIPN) is the most problematic dose-limiting toxicity of oxaliplatin. No treatments have been clinically proven to prevent CIPN. There is a body of evidence that CIPN is caused by cellular oxidative stress. Clinical and preclinical data suggest that the manganese chelate and superoxide dismutase mimetic mangafodipir (MnDPDP) and calmangafodipir ([Ca0.8,Mn0.2]Na3DPDP) are efficacious inhibitors of CIPN and other conditions caused by cellular oxidative stress, without interfering negatively with the tumoricidal activity of chemotherapy.

This is a Phase 3, multicenter, double-blind, placebo-controlled study to establish the efficacious dose of PledOx in prevention of chronic CIPN induced by oxaliplatin.

Patients with metastatic colorectal cancer (mCRC), who are indicated for first-line modified FOLFOX6 (mFOLFOX6) chemotherapy for at least 3 months, without any pre-planned treatment breaks, will be randomized in a 1:1:1 ratio, stratified by region (Asia, non-Asia) and PK sub-study (yes, no), to one of three treatment arms:

* Arm A: PledOx (2 µmol/kg) + mFOLFOX6 chemotherapy
* Arm B: PledOx (5 µmol/kg) + mFOLFOX6 chemotherapy
* Arm C: Placebo + mFOLFOX6 chemotherapy

Before March 2nd., 2020, the Investigational Medicinal Product, (IMP; i.e. PledOx or placebo) was administered by an intravenous infusion on the first day of each chemotherapy (mFOLFOX6) cycle. IMP was not to be administered if mFOLFOX6 was not given to the patient.

If a patient later discontinues oxaliplatin, treatment with 5-FU/folinate may be continued.

The addition of an appropriate biologic therapy (bevacizumab, panitumumab, cetuximab) will be left to the discretion of the Investigator.

As of March 2nd., all patients have to stop IMP but may continue mFOLFOX 6

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form before any study related assessments and willing to follow all study procedures.
* Male or female aged >=18 years.
* Non-resectable metastatic (stage IV) CRC, pathologically confirmed adenocarcinoma of the colon or rectum.
* No prior chemotherapy (within the previous 12 months) and/or biologic/targeted therapy for mCRC.
* Measurable disease according to RECIST 1.1.
* Patient indicated for at least 3 months of oxaliplatin-based chemotherapy (without any pre-planned treatment breaks) and without any clinically observed neurological disorders.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematological parameters: hemoglobin >=100 g/L, absolute neutrophil count (ANC) >=1.5 x 10^9 /L, platelets >=100 x 10^9 /L.
* Adequate renal function: creatinine clearance >50 cc/min using the Cockroft and Gault formula or measured.
* Adequate hepatic function: total bilirubin <=1.5 times the upper limit of normal (ULN) (except in the case of known Gilbert's syndrome); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=3 times ULN (AST and ALT <=5 times ULN in case of liver metastases).
* Baseline blood manganese (Mn) level <2.0 times ULN.
* For patients with a history of diabetes mellitus, HbA1c <=7%.
* Negative pregnancy test for females of child-bearing potential.
* For men and females of childbearing potential, use of adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) while on study drug and for at least 6 months after completion of study therapy.

Exclusion Criteria:

* Any unresolved toxicity by Common Terminology Criteria for Adverse Events Version (CTCAE v4.03) > Grade 1 from previous anti-cancer therapy (including radiotherapy), except alopecia.
* Any grade of neuropathy from any cause.
* Any evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, cardiac, unresolved bowel obstruction, hepatic or renal disease).
* Chronic infection or uncontrolled serious illness causing immunodeficiency.
* Any history of seizures.
* A surgical incision that is not healed.
* Significant hemorrhage (>30 mL/bleeding episode in previous 3 months), hemoptysis (>5 mL fresh blood in previous 4 weeks) or thrombotic event (including transient ischemic attack) in the previous 12 months if the patient is expected to receive anti-VEGF/VEGFR therapy.
* Known hypersensitivity to any of the components of mFOLFOX6 and, if applicable, biological therapies to be used in conjunction with the chemotherapy regimen or any of the excipients of these products.
* History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within 5 years, unless the patient has been disease free for that other malignancy for at least 2 years.
* Known dihydropyrimidine dehydrogenase deficiency.
* Pre-existing neurodegenerative disease (e.g., Parkinson's, Alzheimer's, Huntington's) or neuromuscular disorder (e.g., multiple sclerosis, amyotrophic lateral sclerosis, polio, hereditary neuromuscular disease).
* Major psychiatric disorder (major depression, psychosis), alcohol and/or drug abuse.
* Patients with a history of second or third degree atrioventricular block or a family heredity.
* A history of a genetic or familial neuropathy.
* Treatment with any investigational drug within 30 days prior to randomization.
* Pregnancy, lactation or reluctance to using contraception.
* Any other condition that, in the opinion of the Investigator, places the patient at undue risk.
* Previous exposure to mangafodipir or calmangafodipir.
* Welders, mine workers or other workers in occupations (current or past) where high manganese exposure is likely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Carlsson, MD, Study Director — Chief Medical Officer
Locations (98):
- United States (11):
  - California Cancer Associates, Fresno, California
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Mercy Clinic - Cancer & Hematology, Springfield, Missouri
  - Mercy Clinic Oncology and Hematology, St Louis, Missouri
  - CHI St Francis Cancer Treatment Center, Grand Island, Nebraska
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Monter Cancer Center, Lake Success, New York
  - Montefiore Medical Research, The Bronx, New York
  - Scott & White Vasicek Cancer Treatment Center, Temple, Texas
- Belgium (8):
  - Onze-Lieve-Vrouwziekenuis Aalst, Aalst
  - Imelda GI Clinical Research Center, Bonheiden
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
  - CHU Liège, Liège
  - AZ Sint Maarten, Mechelen
  - AZ Delta, Roeselare
  - CHU UCL Namur - Site Godinne, Yvoir
- Czechia (6):
  - Nemocnice Benesov, Benešov
  - Nemocnice Horovice, Hořovice
  - Nemocnice Na Pleši, Nová Ves pod Pleší
  - General University Hospital, Prague
  - Hospital Na Bulovce, Prague
  - Onkologická Klinika 1. Lf Uk A Tn, Prague
- France (12):
  - CHRU de Brest - Hôpital Morvan, Brest
  - Clinique Pasteur-Lanroze, Brest
  - Centre Hospitalier Départemental de Vendée - Unité de recherche clinique, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Hôpital Edouard Herriot - HCL, Lyon
  - Hôpital Nord Franche-Comté Site du Mittan, Montbéliard
  - Institut de Cancérologie de l'Ouest, Nantes
  - Hopital l'Archet, CHU de Nice, Nice
  - Hôpital Robert Debré, Reims
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Clinique Ste Anne, Strasbourg
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Germany (6):
  - Hämatolgisch-onkologische Praxis Augsburg, Augsburg
  - Onkozentrum Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Onkodok GmbH, Gütersloh
  - Klinikum Neuperlach, München
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (5):
  - Országos Onkológiai Intézet, Budapest
  - Semmelweis Egyetem, Budapest
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelőintézet, Szolnok
- Italy (12):
  - IRCCS Candiolo, Candiolo
  - Oncologia Istituti Ospitalieri, Cremona
  - Irccs Irst, Meldola - FC
  - Azienda Ospedaliero - Universitaria di Modena Policlinico, Modena
  - Hospital San Gerardo, Monza
  - Istituto Nazionale Tumori, Napoli
  - IRCCS Policlinico San Matteo, Pavia
  - Ospedale degli infermi, Ponderano
  - Ospedale S. Maria delle Croci - Ravenna, Ravenna
  - IRCCS azienda Ospedaliera S Maria Nuova, Reggio Emilia
  - San Camillo Forlanini Hospital, Rome
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Japan (12):
  - Osaka International Cancer Institute, Osaka-shi, Osaka, Osaka
  - Fujita Health University Hospital, Aichi
  - Kyushu University Hospital, Fukuoka-shi, Fukuoka
  - Fukuoka University Hospital, Fukuoka-shi, Fukuoka
  - Kansai Rosai Hospital, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Aichi Cancer Center Hospital, Nagoya-shi, Aichi
  - Osaka University Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka-shi, Osaka
  - Sapporo Medical University Hospital, Sapporo-shi, Hokkaido
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital Of JFCR, Tokyo
- South Korea (6):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Dong-A University Hospital, Busan
  - Chonnam National University Hwasun Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (11):
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - L´Hospitalet de Llobregat (Barcelona), Barcelona
  - Vall d'hebron university hospital, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Centro Integral Oncologico Clara Campal, Madrid
  - H.G.U.Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quironsalud Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza
- Taiwan (3):
  - KMUH: Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - CMMC: Chi Mei Medical Center, Tainan
  - NCKUH: National Cheng Kung University Hospital, Tainan
- United Kingdom (5):
  - Royal Marsden Hospital, London
  - North Tyneside General Hospital, North Shields
  - Mount Vernon Cancer Centre, Northwood
  - The Royal Marsden Hospital (Surrey), Sutton
  - York Teaching Hospital, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfeiffer P, Lustberg M, Nasstrom J, Carlsson S, Persson A, Nagahama F, Cavaletti G, Glimelius B, Muro K. Calmangafodipir for Prevention of Oxaliplatin-Induced Peripheral Neuropathy: Two Placebo-Controlled, Randomized Phase 3 Studies (POLAR-A/POLAR-M). JNCI Cancer Spectr. 2022 Nov 1;6(6):pkac075. doi: 10.1093/jncics/pkac075. PMID 36308441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the US, EU and Asia between 2018 and 1 March 2020. The Sponsor placed recruitment/dosing in the POLAR program on hold following interactions with the French regulatory authority and a US clinical hold of the study on 23 January 2020. As of 2 March 2020, no more patients were enrolled or IMP administered. Enrolled patients were followed until the data cut-off date of 31 August 2020 and these patients have been assigned as "completed" in the disposition.
Pre-assignment Details: 386 patients were screened in the 28 days before the start of treatment, 291 were randomised and 285 were treated.
Groups:
- PledOx (2 µmol/kg): Calmangafodipir (2 µmol/kg) on day 1 every two weeks to patients as an intravenous infusion, combined with mFOLFOX6 chemotherapy.
  Calmangafodipir (2 µmol/kg): Solution in 20 mL single dose glass vial
- PledOx (5 µmol/kg): Calmangafodipir (5 µmol/kg) on day 1 every two weeks to patients as an intravenous infusion, combined with mFOLFOX6 chemotherapy.
  Calmangafodipir (5 µmol/kg): Solution in 20 mL single dose glass vial
- Placebo: Placebo will be given to patients as an intravenous infusion, on top of mFOLFOX6 chemotherapy.
  Placebo: Solution in 20 mL single dose glass vial
Period: Overall Study
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Started | 97 | 96 | 98
Treated | 96 | 93 | 96
Completed | 66 | 70 | 69
Not Completed | 31 | 26 | 29
Not completed — Death | 9 | 9 | 16
Not completed — Withdrawal by Subject | 8 | 6 | 4
Not completed — Study terminated by Sponsor | 3 | 5 | 4
Not completed — Not reported | 2 | 4 | 5
Not completed — Progressive disease | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Site terminated by Sponsor | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisting of all randomized patients who received at least one dose of IMP. Patients were analyzed according to the study treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo | Total
Number analyzed (Participants) | 96 | 93 | 96 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.5) | 62.9 (9.6) | 61.6 (12.4) | 62.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 40 | 119
  Male | 60 | 50 | 56 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 41 | 40 | 39 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 49 | 45 | 51 | 145
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 5 | 18
Body Mass Index [Median (Full Range); unit: kg/m^2] | 23.60 [16.5 to 35.3] | 24.20 [17.4 to 40.3] | 24.00 [16.5 to 32.8] | 24.00 [16.5 to 40.3]
ECOG performance status [Count of Participants; unit: Participants] — The ECOG performance scale is a six point functional scale (0 to 5) rating the extent of effect on daily living with higher scores representing a worse outcome. A score 0 represents "fully active, able to carry on all pre-disease performance without restriction" and a score 1 represents "restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work".
  Participants
    0 | 65 | 62 | 53 | 180
    1 | 31 | 31 | 41 | 103
    Unknown | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Moderate or Severe Chronic Chemotherapy Induced Peripheral Neuropathy (CIPN)
Description: Percentage of patients (with moderate or severe chronic CIPN) scoring 3 or 4 in at least 1 of the first 4 items of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-13-item subscale (FACT/GOG-NTX-13; i.e., FACT/GOG-NTX-4) 9 months after the first dose of IMP (i.e. PledOx or placebo administered on Day 1, Cycle 1 of mFOLFOX6 chemotherapy). The FACT/GOG-13 questionnaire includes 13 items that measure the severity and impact of symptoms of neurotoxicity over the past 7 days. Patients rate each item as 0 ("not at all"), 1 (" a little bit"), 2 ("somewhat"), 3 ("quite a bit") or 4 ("very much"). These 13 items are summed to create a total score, ranging from 0 to 52, with a higher score representing a worse outcome. The FACT/GOG-NTX-4 is a 4 item subscale targeting numbness, tingling or discomfort in hands and/or feet.
Time Frame: 9 months
Population: Modified ITT (mITT) analysis set including patients that fulfilled at least one of the following criteria:
  * the patient was randomized prior to 1 Dec 2019 (i.e. the patient was eligible for at least 3 months of IMP) and had at least one post-baseline assessment for efficacy, or
  * the 3 month Assessment Visit occurred prior to 1 Mar 2020, or
  * the patient received the 6th cycle of IMP after 1 Mar 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 54 | 55 | 57
Participants | 31 | 27 | 25
Statistical Analysis 1: Comparison: PledOx (2 µmol/kg) vs Placebo; Cochran-Mantel-Haenszel estimate of the common relative risk of moderate to severe CIPN; Test type: Superiority; p = 0.2266, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.3842, 95% CI 2-sided [0.8172 to 2.3446]
Statistical Analysis 2: Comparison: PledOx (5 µmol/kg) vs Placebo; Cochran-Mantel-Haenszel estimate of the common relative risk of moderate to severe CIPN; Test type: Superiority; p = 0.7434, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.0951, 95% CI 2-sided [0.6356 to 1.8870]

2. Secondary Outcome: Mild, Moderate or Severe Chronic Chemotherapy Induced Peripheral Neuropathy (CIPN)
Description: Percentage of patients (with mild, moderate or severe chronic CIPN) scoring 2, 3 or 4 in at least 1 of the first 4 items of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-13-item subscale (FACT/GOG-NTX-13; i.e., FACT/GOG-NTX-4) 9 months after the first dose of IMP (i.e. PledOx or placebo administered on Day 1, Cycle 1 of mFOLFOX6 chemotherapy). The FACT/GOG-13 questionnaire includes 13 items that measure the severity and impact of symptoms of neurotoxicity over the past 7 days. Patients rate each item as 0 ("not at all"), 1 (" a little bit"), 2 ("somewhat"), 3 ("quite a bit") or 4 ("very much"). These 13 items are summed to create a total score, ranging from 0 to 52, with a higher score representing a worse outcome. The FACT/GOG-NTX-4 is a 4 item subscale targeting numbness, tingling or discomfort in hands and/or feet.
Time Frame: 9 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 54 | 55 | 57
Participants | 43 | 40 | 42

3. Secondary Outcome: Sensitivity to Touching Cold Items
Description: Mean change from baseline in sensitivity to touching cold items on day 2, Cycle 4 of mFOLFOX6 chemotherapy, as assessed by the Cold Sensitivity Questionnaire (measuring sensitivity when touching or swallowing cold objects/fluid). 10 point scale from 0 meaning no sensitivity/discomfort at all to 10 meaning sensitivity/discomfort as bad as it can be.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 68 | 66 | 66
Scores on a scale | 3.88 [3.19 to 4.57] | 4.13 [3.43 to 4.82] | 3.41 [2.71 to 4.11]

4. Secondary Outcome: Cumulative Dose of Oxaliplatin During Chemotherapy
Description: Mean cumulative dose of oxaliplatin administered per patient during mFOLFOX6 chemotherapy, 9 months after the first dose of IMP.
Time Frame: 9 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/m^2
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 80 | 78 | 78
mg/m^2 | 780.69 [711.86 to 849.52] | 803.54 [734.01 to 873.07] | 764.52 [694.91 to 834.14]

5. Secondary Outcome: Vibration Sensitivity on the Lateral Malleolus
Description: Mean change from baseline in vibration sense, on the lateral malleolus (left and right), using a graduated tuning fork, at 9 months after the first dose of IMP. When the tuning fork was struck against the ball of the thumb, the base of the tuning fork was placed over the appropriate bony surface (i.e., lateral malleolus left and right) and the patient was asked to indicate the moment when the vibration was no longer detected. The intensity at which the patient no longer detected the vibration is reported on a scale of 0 (minimum score, representing the maximum vibration amplitude) to 8 (maximum score, representing the minimum vibration amplitude)
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 49 | 49 | 51
Scores on a scale | -1.53 (2.06) | -1.61 (2.09) | -1.36 (1.68)

6. Secondary Outcome: Worst Pain in Hands or Feet
Description: Mean change from baseline in worst pain in hands or feet in the past week, using the Pain Assessment (Numerical Rating Scale (NRS)), at 9 months after the first dose of IMP. The NRS is a 10 point scale with 0 as no pain at all and 10 as pain as bad as you can imagine and evaluates the intensity of pain in hands and feet during the past week. A higher value means worse outcome.
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 51 | 52 | 54
Scores on a scale | 2.19 [1.37 to 3.01] | 1.58 [0.76 to 2.39] | 1.92 [1.12 to 2.72]

7. Secondary Outcome: Functional Impairment (in the Non-dominant Hand)
Description: Mean change from baseline in the time to complete the grooved Pegboard with the non-dominant hand, at 9 months after the first dose of IMP.
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 45 | 47 | 50
seconds | 9.68 [-3.07 to 22.44] | 14.24 [1.72 to 26.75] | 12.01 [-0.07 to 24.09]

8. Secondary Outcome: Overall Response Rate (ORR)
Description: Percentage of patients with an overall response (complete response or partial response) according to RECIST v1.1 for target lesions and assessed by CT (preferred) or MRI. Complete response=disappearance of all target lesions; partial response >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 12, 15 and 18 months
Population: The safety analysis set consisting of all randomized patients who received at least one dose of IMP. The overall number analyzed represents the total in the safety population treated at the start of the study. ORR was assessed throughout the study when varying numbers of patients in each group remained on study
Measure: Count of Participants; unit: Participants
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 96 | 93 | 96
Participants
  Month 12: number analyzed (Participants) | 41 | 44 | 39
  Month 12: Missing | 22 | 19 | 19
  Month 12: No | 6 | 13 | 12
  Month 12: Yes | 13 | 12 | 8
  Month 15: number analyzed (Participants) | 22 | 23 | 12
  Month 15: Missing | 9 | 14 | 7
  Month 15: No | 7 | 7 | 3
  Month 15: Yes | 6 | 2 | 2
  Month 18: number analyzed (Participants) | 4 | 6 | 2
  Month 18: Missing | 1 | 3 | 1
  Month 18: No | 2 | 3 | 0
  Month 18: Yes | 1 | 0 | 1

9. Secondary Outcome: Progression-free Survival (PFS)
Description: Patients with progression-free survival
Time Frame: Analyses at 12 and 24 months were planned; the analysis was performed once based on available data at cut-off 31 August 2020 as the study was terminated early by the Sponsor
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 95 | 93 | 95
participants | 40 | 36 | 36

10. Secondary Outcome: Overall Survival (OS)
Description: Patients with overall survival
Time Frame: An analysis at 36 months was planned. The analysis was performed based on available data at cut-off 31 August 2020 as the study was terminated early by the Sponsor
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 95 | 93 | 95
participants | 9 | 9 | 16

ADVERSE EVENTS:
Time Frame: From screening until 30 days after the end of treatment visit which occurred after up to 6 months of treatment
Arm/Group | PledOx (2 µmol/kg) | PledOx (5 µmol/kg) | Placebo
All-Cause Mortality (participants affected / at risk) | 9/96 | 9/93 | 16/96
Serious Adverse Events (participants affected / at risk) | 27/96 | 21/93 | 24/96
Other Adverse Events (participants affected / at risk) | 93/96 | 91/93 | 95/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PledOx (2 µmol/kg) (N=96) | PledOx (5 µmol/kg) (N=93) | Placebo (N=96)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (2)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PledOx (2 µmol/kg) (N=96) | PledOx (5 µmol/kg) (N=93) | Placebo (N=96)
Anaemia (Blood and lymphatic system disorders) | 11 (17) | 8 (15) | 14 (23)
Leukopenia (Blood and lymphatic system disorders) | 12 (29) | 10 (22) | 14 (26)
Neutropenia (Blood and lymphatic system disorders) | 40 (91) | 48 (97) | 37 (90)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (26) | 16 (28) | 16 (36)
Abdominal pain (Gastrointestinal disorders) | 16 (21) | 14 (21) | 16 (18)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (5) | 5 (6)
Constipation (Gastrointestinal disorders) | 24 (26) | 15 (17) | 14 (19)
Diarrhoea (Gastrointestinal disorders) | 32 (56) | 27 (27) | 41 (68)
Dyspesia (Gastrointestinal disorders) | 8 (10) | 6 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 34 (67) | 42 (69) | 47 (82)
Stomatitis (Gastrointestinal disorders) | 29 (39) | 24 (41) | 29 (43)
Vomiting (Gastrointestinal disorders) | 11 (24) | 16 (32) | 20 (30)
Asthenia (General disorders) | 14 (23) | 17 (47) | 21 (41)
Fatigue (General disorders) | 25 (38) | 23 (33) | 23 (35)
Malaise (General disorders) | 6 (6) | 4 (5) | 9 (10)
Oedema peripheral (General disorders) | 6 (8) | 3 (3) | 4 (5)
Pyrexia (General disorders) | 12 (15) | 8 (11) | 9 (10)
Drug hypersensitivity (Immune system disorders) | 5 (6) | 2 (2) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (5) | 4 (5) | 5 (5)
Paronychia (Infections and infestations) | 2 (3) | 7 (8) | 8 (9)
Alanine aminotransferase increased (Investigations) | 5 (5) | 7 (8) | 8 (16)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 7 (8) | 7 (16)
Decreased appetite (Metabolism and nutrition disorders) | 30 (47) | 26 (33) | 27 (42)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (3) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 7 (11) | 9 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 7 (8) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5) | 6 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (9) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 10 (13)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5) | 6 (8)
Dysgeusia (Nervous system disorders) | 16 (18) | 20 (23) | 21 (24)
Headache (Nervous system disorders) | 7 (10) | 7 (7) | 5 (6)
Neuropathy peripheral (Nervous system disorders) | 32 (89) | 33 (84) | 36 (74)
Paraesthesia (Nervous system disorders) | 17 (26) | 15 (25) | 18 (35)
Peripheral sensory neuropathy (Nervous system disorders) | 42 (86) | 40 (79) | 42 (97)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3) | 5 (5)
Proteinuria (Renal and urinary disorders) | 5 (6) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (18) | 14 (15) | 9 (13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 3 (6) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 11 (14) | 13 (13)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 (15) | 7 (8) | 10 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9) | 11 (11) | 4 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (10) | 4 (6) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (13) | 19 (30) | 14 (18)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (7) | 1 (1)
Hypertension (Vascular disorders) | 12 (12) | 11 (16) | 12 (16)
Weight decreased (Investigations) | 10 (12) | 4 (4) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03654729/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03654729/SAP_001.pdf